CLINICAL TRIAL: NCT03325595
Title: A Phase 1, Single Center, Double-blind, Placebo-controlled, Dose Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Effects of Single Oral Doses of AEF0117 in Healthy Male and Female Subjects
Brief Title: Single Ascending Dose to Study the Safety, Tolerability, PK and PD Effects of AEF0117
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AEF0117-101; R01DA038875 (NIH)
Record Dates: First submitted 2017-10-11; First posted 2017-10-30 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study. Subjects and investigator will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: AEF0117 (Active Comparator): Subjects in Cohorts 1 through 4 receive active treatments. Subjects in Cohorts 1 through 4 will receive a single dose of 0.2, 0.6, 2 and 6mg respectively of AEF0117 on Day1.
  Interventions: Drug: AEF0117
- Placebo Comparator: Placebo (Placebo Comparator): Subjects in Cohorts 1 through 4 will be randomly assigned in an 6:2 allocation to receive active or placebo treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AEF0117 — 0.2, 0.6, 2, or 6mg of AEF0117
  Arms: Experimental: AEF0117
Drug: Placebo — Matching capsule placebo
  Arms: Placebo Comparator: Placebo

SUMMARY:
The study is designed to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of escalating single oral doses of AEF0117 in healthy adult male and female subjects.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of escalating single oral doses of AEF0117 in healthy adult male and female subjects. This will be a single center study in healthy adult male and female subjects. The study design will be a double-blind, randomized, placebo-controlled, single period, parallel group, single dose escalation with AEF0117.

Four dose levels are planned for the study with 8 subjects (6 active and 2 placebo, 3:1 ratio) per dose level:

Dose Level I - 0.2 mg single oral dose of AEF0117 given on the morning of Day 1 Dose Level II - 0.6 mg single oral dose of AEF0117given on the morning of Day 1 Dose Level III - 2 mg single oral dose of AEF0117 given on the morning of Day 1 Dose Level IV - 6 mg single oral dose of AEF0117 given on the morning of Day 1 The planned dose escalation schema may be amended based on the emerging PK and safety data. Each subject will participate in only one dose group.

In each dosing cohort, 2 sentinel subjects (randomized 1 AEF0117: 1placebo) will be dosed and observed for safety monitoring for 24 hours prior to initiating dosing in the remaining 6 subjects (randomized 5 AEF0117: 1 placebo).

The first cohort will be administered 0.2mg. Administration of AEF0117 to the subsequent dose cohorts,0.6 mg(Cohort II), 2 mg (Cohort III), and 6 mg (Cohort IV) doses should not occur before participants in the previous dose cohort have been treated and data i.e. safety results from those participants are reviewed in accordance with the protocol.

Serial blood sample collections will be performed for 144 hours after dose administration for PK analysis, and for 48 hours after dose administration for PD analysis.

Subjects will be admitted to the research clinic at midday prior to dosing (Day -1) and remain in-house until Day 8. Randomized subjects will receive a single dose of AEF0117 on Day 1. PK samples and safety assessments will be performed pre-dose and at different times post dose. Safety monitoring (physical examinations, vital sign measurement, 12-lead electrocardiograms [ECGs], clinical safety laboratory tests, and adverse event monitoring) will be performed throughout the study. Psychometrics (Bond & Lader VAS, ARCI, POMS) and C-SSRS tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Be a healthy, non-smoking or smoking (<10 cigarettes per day) male of any race, at least 18 years old and no more than 55 years old, inclusive. As the effect of the study drug on sperm is still unknown, male subjects should refrain from donating sperm or plan a pregnancy with their partner throughout the study and after 90 days, and must report immediately to the study doctor if its partner becomes pregnant during the study and after 90 days. The male subject will have to use double-barrier contraceptive methods: male condoms and spermicide.
2. Be a healthy, non-smoking or smoking (<10 cigarettes per day) female of non-child-bearing potential between 18 years of age and 55 years of age, inclusive. Females may be accepted if they are documented to be surgically sterile (e.g., hysterectomy, tubal ligation) or post-menopausal [amenorrhea >1 year and FSH >25.8mlU/mL, cut off from Labcorp] with a negative pregnancy test. At least 30% of female.
3. Have a body weight ≥50 kg, with a body mass index (BMI) calculated as weight in kg/(height in m)2 from 18 to 30 kg/m2 (inclusive) at screening.
4. Have no significant diseases in the medical history and no clinically significant findings on physical examination including ECG, BP, HR, RR, temperature, C-SSRS test. Routine laboratory values should be within normal ranges or considered as NCS by the investigator. The Non Clinical Significant nature of the deviation will result from the integration of a full clinical examination with physical examination and lab tests in that contest by a certified physician.
5. Be informed of the nature of the study and provide written informed consent.
6. Be legally competent and able to communicate effectively with study personnel.

Exclusion Criteria:

1. Allergies to the Investigational Medicinal Product (IMP) or placebo and its excipients and known allergies to pregnenolone or its matching placebo or its ingredient
2. Acute signs of intoxication at screening or baseline assessment due to opiates or any type of stimulants, causing cognitive impairments
3. Severe learning disability, brain damage or pervasive developmental disorder ( as this may affect one of the end point that is being targeted)
4. Any disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems.
5. Have abnormal baseline values for the steroid hormones: cortisol, testosterone, estradiol and progesterone in accordance to their reproductive status (for example but not limited to surgical sterile or post-menopausal).
6. A history of alcoholism or drug addiction within the past 2 years, recent use (in the last month) of any recreational drugs, or positive results from a urine screen for substances of abuse or from an alcohol breath test.
7. A history of or current serious mental illness including active or recent suicidal ideation, severe psychological distress (e.g., active suicidal plans, psychosis, debilitating panic disorder) or/and an abnormal C-SSRS result.
8. A history of difficulty donating blood or inadequate venous access.
9. The donation of blood or plasma within 30 days prior to receiving study medication or received any blood and plasma for medical/surgical reasons or intention to donate blood or plasma within one month after receiving the study drug.
10. A positive hepatitis screen that tests for both hepatitis B surface antigen (HBsAg) and antibody to hepatitis C (HCV).
11. A positive test result for HIV antibody by enzyme immunoassay which is confirmed by Western immunoblot.
12. Ingestion of an investigational drug or product, or participation in a drug study within a period of 30 days prior to receiving study medication (for investigational drugs with an elimination half-life greater than 10 days, this will be extended to 60 days).
13. Use of any prescription or over-the-counter (OTC) drug therapy, including herbal, homeopathic, vitamins, minerals and nutritional supplements, bodybuilding supplements unapproved by the sponsor, within 2 weeks prior to receiving the study medication (for drugs with an elimination half-life greater than 10 days, this will be extended to 60 days). The use of any food supplement or body cream containing pregnenolone or any other steroid including phytosteroids.
14. Use of a drug therapy known to induce or inhibit hepatic drug metabolism within 30 days prior to receiving study medication or during the study.
15. Use of psychoactive and/or psychotropic medication (including sedative, antidepressant and antipsychotics), or medication that alters the hypothalamic pituitary adrenal (HPA) Axis functioning and any medications that alter heart rate or skin conductance monitoring.
16. Unable to follow the restrictions outlined in the protocol.
17. Legal status that would interfere with participation.
18. Employed by the contract research organization (CRO) or are family members of the staff at the CRO.
19. Previous participation in a cohort for any dose level of AEF0117.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent AEs and SAEs as assessed by vital signs | 168 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in vital signs
Incidence of treatment-emergent AEs and SAEs as assessed by ECGs | 168 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in ECGs
Incidence of treatment-emergent AEs and SAEs as assessed by clinical laboratory values | 168 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in clinical laboratory values from blood and urine samples.
Incidence of treatment-emergent AEs and SAEs as assessed by psychometric tests | 36 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in psychometric tests (Bond and Lader VAS, ARCI, POMS) and C-SSRS test.

SECONDARY OUTCOMES:
Pharmacokinetics of escalating single oral doses of AEF0117 | 144 hours from dosing
  Peak Plasma Concentration (Cmax) induced by a single dose of AEF0117will be determined based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating single oral doses of AEF0117 | 144 hours from dosing
  Lowest Peak Plasma (Cmin) induced by a single dose of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating single oral doses of AEF0117 | 144 hours from dosing
  Time to maximum plasma concentration (tmax) of a single dose of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating single oral doses of AEF0117 | 144 hours from dosing
  Terminal elimination half-life (t1/2) based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating single oral doses of AEF0117 | 144 hours from dosing
  Time to last measurable plasma concentration (tlast) based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacokinetics of escalating single oral doses of AEF0117 | 144 hours from dosing
  Area under the plasma concentration versus time curve from time 0 (AUC0-t) based on serial blood sample collections and plasma AEF0117 concentration.
Pharmacodynamics of escalating single oral doses of AEF0117 | 48 hours from dosing
  Peak Plasma Concentration (Cmax) induced by a single dose of AEF0117 on plasma pregnenolone, 17-OH-pregnenolone, DHEA, allopregnanolone, testosterone and endocannabinoids (AEA and 2AG) and serum estradiol, progesterone and cortisol concentrations.
Pharmacodynamics of escalating single oral doses of AEF0117 | 48 hours from dosing
  Lowest Peak Plasma (Cmin) induced by a single dose of AEF0117 on plasma pregnenolone, 17-OH-pregnenolone, DHEA, allopregnanolone, testosterone and endocannabinoids (AEA and 2AG) and serum estradiol, progesterone and cortisol concentrations.
Pharmacodynamics of escalating single oral doses of AEF0117 | 48 hours from dosing
  Time to maximum plasma concentration (tmax) of a single dose of AEF0117 on plasma pregnenolone, 17-OH-pregnenolone, DHEA, allopregnanolone, testosterone and endocannabinoids (AEA and 2AG) and serum estradiol, progesterone and cortisol concentrations.
Pharmacodynamics of escalating single oral doses of AEF0117 | 48 hours from dosing
  Area under the plasma concentration versus time curve from time 0 (AUC0-t) of a single dose of AEF0117 on plasma pregnenolone, 17-OH-pregnenolone, DHEA, allopregnanolone, testosterone and endocannabinoids (AEA and 2AG) and serum estradiol, progesterone and cortisol concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dobrow, MD, Principal Investigator — Biotrial Inc.
Locations (1):
- Biotrial Inc, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haney M, Vallee M, Fabre S, Collins Reed S, Zanese M, Campistron G, Arout CA, Foltin RW, Cooper ZD, Kearney-Ramos T, Metna M, Justinova Z, Schindler C, Hebert-Chatelain E, Bellocchio L, Cathala A, Bari A, Serrat R, Finlay DB, Caraci F, Redon B, Martin-Garcia E, Busquets-Garcia A, Matias I, Levin FR, Felpin FX, Simon N, Cota D, Spampinato U, Maldonado R, Shaham Y, Glass M, Thomsen LL, Mengel H, Marsicano G, Monlezun S, Revest JM, Piazza PV. Signaling-specific inhibition of the CB1 receptor for cannabis use disorder: phase 1 and phase 2a randomized trials. Nat Med. 2023 Jun;29(6):1487-1499. doi: 10.1038/s41591-023-02381-w. Epub 2023 Jun 8. PMID 37291212